CLINICAL TRIAL: NCT03500965
Title: Pictorial Warning Labels and Memory for Relative and Absolute Cigarette Health-risk Information Over Time in Teens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Ellen Peters, Professor, Ohio State University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: P50CA180908A2a-T; P50CA180908 (NIH)
Record Dates: First submitted 2018-02-14; First posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Smoking Cessation; Smoking, Cigarette
Keywords: pictorial warning labels; risk knowledge; emotion; memory; risk perceptions; quit intentions
MeSH Terms: conditions — Smoking Cessation; Cigarette Smoking | interventions — Numbers Needed To Treat; Risk

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Text-only PWL, absol risk (Experimental): Exposure to FDA-mandated warning labels, without a graphic image, accompanied by risk information about smoker's risk of a smoking-related disease
  Interventions: Behavioral: text-only PWL; Behavioral: absolute risk
- text-only PWL, relative risk (Experimental): Exposure to FDA-mandated warning labels, without a graphic image, accompanied by risk information about smoker's risk and non-smoker's risk of a smoking-related disease
  Interventions: Behavioral: text-only PWL; Behavioral: relative risk
- graphic PWL, absol risk (Experimental): Exposure to FDA-mandated warning labels, paired with a graphic image, accompanied by risk information about smoker's risk of a smoking-related disease
  Interventions: Behavioral: graphic PWL; Behavioral: absolute risk
- graphic PWL, relative risk (Experimental): Exposure to FDA-mandated warning labels, paired with a graphic image, accompanied by risk information about smoker's risk and non-smoker's risk of a smoking-related disease
  Interventions: Behavioral: graphic PWL; Behavioral: relative risk

INTERVENTIONS:
Behavioral: text-only PWL — control condition (no image)
  Arms: Text-only PWL, absol risk; text-only PWL, relative risk
Behavioral: graphic PWL — pictorial warning
  Arms: graphic PWL, absol risk; graphic PWL, relative risk
Behavioral: absolute risk — Percentage risk information for smoking-related diseases for smokers
  Arms: Text-only PWL, absol risk; graphic PWL, absol risk
Behavioral: relative risk — Percentage risk information for smoking-related diseases for smokers and non-smokers
  Arms: graphic PWL, relative risk; text-only PWL, relative risk

SUMMARY:
Pictorial cigarette warning labels (PWLs) are thought to increase risk knowledge, but experimental research has not examined PWLs' longer term effects on memory for health risks. In this study, teens who have experimented with smoking or are considered vulnerable to smoking are repeatedly exposed to text-only vs. graphic warning labels paired with numeric risk information. This study will allow us to assess the extent to which reactions to warnings remain consistent over time and influence future smoking intentions. We will also assess the impact of graphic images on memory for smoking risk information presented in absolute and (a smokers lifetime risk of getting a smoking related disease), or relative (a smokers risk of getting a smoking related disease, compared to the risk of non-smokers) formats.

ELIGIBILITY:
Inclusion Criteria:

* have ever tried smoking
* report vulnerability to smoking (i.e., report that they might smoke in the next year or would try a cigarette if a friend offered one)
* parents give permission to participate

Exclusion Criteria:

* not vulnerable to smoking (i.e., report they will definitely not smoke a cigarette in the next year and definitely would not try a cigarette if one was offered
* parents do not provide permission to participate

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 422 (Actual)
Dates: Start 2016-05-25 (Actual); Primary Completion 2018-01-09 (Actual); Study Completion 2018-01-09 (Actual)

PRIMARY OUTCOMES:
numeric risk recognition | measured immediately following last exposure
  Participants answered one multiple choice question about the numeric risk for smokers for each label (e.g., ____% of smokers die before age 85). For each question, there were four decoy responses.

SECONDARY OUTCOMES:
numeric risk recognition | measured after 6-week delay
  Participants answered one multiple choice question about the numeric risk for smokers for each label (e.g., ____% of smokers die before age 85). For each question, there were four decoy responses.
relative risk recognition | measured immediately following last exposure
  Participants answered one multiple choice question about the numeric risk for smokers vs. nonsmokers for each health risk (e.g., a smoker is ____ as likely to die from heart disease as a nonsmoker). For each question, there were three decoy responses (e.g., for heart disease, response options were: "about as likely," "1.75 times," "4.1 times," "10.4 times").
relative risk recognition | measured after 6-week delay
  Participants answered one multiple choice question about the numeric risk for smokers vs. nonsmokers for each health risk (e.g., a smoker is ____ as likely to die from heart disease as a nonsmoker). For each question, there were three decoy responses (e.g., for heart disease, response options were: "about as likely," "1.75 times," "4.1 times," "10.4 times").
smoking risk perceptions | measured immediately following last exposure
  Participants completed several scale items about how much risk they perceived smoking posed to them (e.g., "If a person smokes at your age, how likely are they to get a life-threatening illness from smoking someday ?" [1=very unlikely; 5=extremely likely])
smoking risk perceptions | measured after 6-week delay
  Participants completed several scale items about how much risk they perceived smoking posed to them (e.g., "If a person smokes at your age, how likely are they to get a life-threatening illness from smoking someday ?" [1=very unlikely; 5=extremely likely])
quit intentions (for next 30 days) | measured immediately following last exposure
  Participants intentions to quit smoking; self-reported likelihood of smoking "within the next 30 days" (-3 = very unlikely, 3 = very likely)
  (only for those teens who currently smoked)
quit intentions (for next 30 days) | measured after 6-week delay
  Participants intentions to quit smoking; self-reported likelihood of smoking "within the next 30 days" (-3 = very unlikely, 3 = very likely)
  (only for those teens who currently smoked)
quit intentions (for next year) | measured immediately following last exposure
  Participants intentions to quit smoking; self-reported likelihood of smoking "within the next year" (-3 = very unlikely, 3 = very likely)
  only for those teens who currently smoked
quit intentions (for next year) | measured after 6-week delay
  Participants intentions to quit smoking; self-reported likelihood of smoking "within the next year" (-3 = very unlikely, 3 = very likely)
  only for those teens who currently smoked
risk recognition | measured immediately following last exposure
  Participants were given a list of 9 warnings and asked to select which ones they'd been previously exposed to
risk recognition | measured after 6-week delay
  Participants were given a list of 9 warnings and asked to select which ones they'd been previously exposed to
feelings about smoking | measured immediately following last exposure
  Participants completed several scale items about their feelings towards smoking (e.g., "How good or bad do you feel about smoking?" -2=very bad; +2=very good; "How much do you feel confused about the harms vs. benefits of smoking?" 0=not at all confused; 4=very confused)
feelings about smoking | measured after 6-week delay
  Participants completed several scale items about their feelings towards smoking (e.g., "How good or bad do you feel about smoking?" -2=very bad; +2=very good; "How much do you feel confused about the harms vs. benefits of smoking?" 0=not at all confused; 4=very confused)